CLINICAL TRIAL: NCT05869617
Title: Determining the Effectiveness of Aquatic Exercise in Comparison to Land-based Exercise for Canadian Military Veterans Experiencing Chronic Lower Extremity Musculoskeletal Pain: A Feasibility Study for a Randomized Clinical Trial
Brief Title: Aquatic Exercise for Veterans in Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Nicholas Held (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor-Investigator, Dr. Nicholas Held, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6036919
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain
Keywords: Exercise; military Veterans
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome questionnaires are completed prior to participants being allocated to treatment groups. Unable to blind participants as it is obvious that they will be exercise on land or in water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Land-based exercise (Active Comparator): Traditional active exercise in an land-based setting (i.e., gym) has been shown to be effective in improving chronic pain management.
  Interventions: Other: Land-based Exercise
- Aquatic exercise (Experimental): Exercise completed in a therapy pool with warm water that is matched to the active comparator.
  Interventions: Other: Aquatic exercise

INTERVENTIONS:
Other: Aquatic exercise — Participants in the aquatic therapy group will receive aquatic therapy in a HydroWorx aquatic therapy pool at Hydrathletics.
  In the aquatic therapy group the 20 minutes of aerobic exercise at each visit will involve walking on an underwater treadmill. The intensity of the walking will be determined by the participant at self-selected intensities that are not perceived to cause a lasting increase in pain for one hour after the exercise session.
  The 20 minutes of strengthening exercise will focus on movement patterns that simulate common daily functional activities. Initial intensity of exercises will be determined in collaboration between the health professional and patient by testing the intensity of the exercise that allows the participant to perform 8 repetitions without experiencing a lasting increased in pain. Exercise intensity will be increased weekly by either increasing the number of repetitions or increasing resistance.
  Arms: Aquatic exercise
Other: Land-based Exercise — Traditional land-based training will take place the Hydrathletics gym with similar exercises provided to the aquatic therapy group.
  The aerobic exercise for the land-based therapy group will be 20 minutes of treadmill walking. The intensity will be determined by the participant at self-selected intensities that are not perceived to cause a lasting increase in pain for one hour after the exercise session.
  The 20 minutes of strengthening exercise will focus on similar movement patterns to the aquatic therapy group to simulate common daily functional activities. Initial intensity of exercises will be determined in collaboration between the health professional and patient by testing the intensity of the exercise that allows the participant to perform 8 repetitions without experiencing a lasting increased in pain. Exercise intensity will be increased weekly by either increasing the number of repetitions or the resistance used for the exercise.
  Arms: Land-based exercise

SUMMARY:
This trial is to show the feasibility of administering a randomized clinical trial that determines the effectiveness of aquatic exercise compared to land-based exercise of military Veterans who have chronic pain.

DETAILED DESCRIPTION:
As of March 31, 2020, Veterans Affairs Canada estimated the total Veteran population in Canada to be 629,300. It has been reported that 41 percent of Veterans experience constant pain or discomfort, which is close to double the 22 percent reported by the Canadian population. Pain is a complex phenomenon that involves biological, psychological, and social determinants and impacts. Evidence suggests Veterans have unique pain management needs and evaluation of interventions is urgently needed to address the complex needs of Canadian Military Veterans living with chronic pain.

Aquatic therapy is a possible treatment option that may improve outcomes in military Veterans with chronic pain. Aquatic therapy has previously been shown to decrease pain, improve function or disability, increase quality of life, and improve health-related fitness measures . Most of the research showing effectiveness of aquatic therapy for musculoskeletal pain conditions has involved comparing aquatic therapy to a control group; however, a control group does not accurately reflect current best practice for people with lower extremity musculoskeletal pain. Clinical practice guidelines suggest physical activity and exercise interventions as first-line treatment for people with lower extremity musculoskeletal pain, but do not provide direction on what type of exercise is most effective for people with lower extremity pain. Building on existing research by comparing aquatic therapy to a land-based exercise comparison will provide a more robust evaluation of the effectiveness to inform clinical practice guidelines. Additionally, given their unique health needs, there is a need for evidence specific to the military Veteran population.

To date, there have been eight randomized clinical trials comparing aquatic exercise to land-based exercise on function or disability for people with lower extremity musculoskeletal pain. While meta-analyses reveal no difference between these two groups in pain, function, and quality of life, this body of research is limited by small sample sizes and risks of bias, making it difficult to draw conclusions and apply the evidence of effectiveness in practice. There are opportunities to improve rigor by reducing the risk of bias (e.g., most studies did not describe allocation concealment) and conducting a fully powered trial. Additionally, important differences between groups in satisfaction of participants and a gap in terms of understanding the experiences are emerging. Further research on the experiences and perspectives of participants is needed. Most importantly, there have been no studies on the effectiveness or experiences of aquatic therapy among Canadian Military Veterans living with pain. Given the unique needs of this population, evidence specific to this group is needed in order to inform service delivery.

Prior to conducting a fully powered trial, there is a need for a pilot study to determine the feasibility of carrying out the interventions and trial procedures. Primarily, the ability to recruit Canadian Military Veterans who live with chronic pain into the study and to determine if participants have the opportunity to book and attend two sessions per week for eight weeks.

Objectives:

1. Determine feasibility of trial methods, including patient recruitment rate, assessment procedures, and attrition.
2. Determine the feasibility of implementing the aquatic exercise and land-based exercise interventions as designed.
3. Explore the perspectives of patients and health professionals related to the acceptability of the interventions and trial methods, barriers, facilitators and strategies for implementation; and perceived impact on clinic processes and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Canadian Armed Forces Veteran
* Living with lower-extremity musculoskeletal chronic pain (>12 weeks)

Exclusion Criteria:

* Pain of < 12 weeks duration
* cancer-related pain and pain suspected to be associated with a degenerative neurological condition
* surgery or fracture in the last 6 months
* medical contraindications to exercise (e.g., recent myocardial infarction, acute heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 1 year
  participants recruited per week.
Retention rate | Through study completion, an average of 1 year
  percentage of participants who complete the scheduled follow-up assessments at each time point.
Outcome measure completion rate | Through study completion, an average of 1 year
  percentage of items completed across all outcome measures at all time points.
Treatment fidelity | Through study completion, an average of 1 year
  using a treatment fidelity checklist, as describe below, we will consider how often a practitioner adheres to the recommended exercises and if the participants complete all exercises in a session.
Treatment adherence | Through the length of the intervention, completed at 8 weeks
  measured based on attendance through the treatment fidelity checklist. In an 8-week period, participants will be asked to attend 16 sessions which will be confirmed by the practitioner handing in the fidelity checklist to the study team after each session.

SECONDARY OUTCOMES:
Physical function | Pre-intervention (0 weeks), post-intervention (8 weeks) and follow-up (20 weeks).
  Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS has previously been shown to be reliable, and construct validity has been supported by comparison with the SF-36. A score is provided for each of the 20 activities from 0 (extreme difficulty or unable to perform activity) to 4 (no difficulty). LEFS is scored by summating all points for all activities to equate a minimum score of zero and a maximum score of 80. The lower the score, the greater the associated disability. A minimal detectable change of 9 points has been reported for LEFS.
Pain severity | Pre-intervention (0 weeks), post-intervention (8 weeks) and follow-up (20 weeks).
  Brief Pain Inventory (BPI) is a questionnaire developed to assess the severity of pain and pain interference. The severity index will be used to determine pain levels at the three time points of interest. The BPI has been validated previously for the assessment of pain severity, including musculoskeletal pain. Mean pain severity is scored by self-reporting the average pain on a 10-point scale from "no pain" to "pain as bad as you can imagine".
Pain interference | Pre-intervention (0 weeks), post-intervention (8 weeks) and follow-up (20 weeks).
  the Brief Pain Inventory (BPI) interference index will be used to assess pain interference. The BPI -Pain interference index measures how much pain interferes with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations to others, and sleep. Each of the seven questions is scored on a scale from 0-10 with higher scores representing more interference. Pain interference is scored as the mean of the seven interference items. Scores in these seven areas can be categorized as affective interference (enjoyment with life, mood, and relations to others) and activity interference (general activity, walking, work, and sleep) subscales.
Health-related quality of life | Pre-intervention (0 weeks), post-intervention (8 weeks) and follow-up (20 weeks).
  The EuroQol EQ-5D-5L is a validated, self-reporting tool used to assess quality of life based on five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Under each dimension, participants check a box that best indicates the level of problems they have within that dimension. Each box is coded from 1 (no problem) to 5 (severe problems). Additionally, participants complete a 100-point visual analog scale on their overall health for the day.
Sleep quality | Pre-intervention (0 weeks), post-intervention (8 weeks) and follow-up (20 weeks).
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality and disturbance retrospectively over a 1-month period using self-reports. PSQI scores are moderately to highly correlated with measures of sleep quality and sleep problems, and poorly correlated with unrelated constructs. Individuals with sleep problems, poor sleep quality, and sleep restlessness score significantly higher PSQI scores in comparison to individuals without such problems. The PSQI includes 19 self-rated questions that are combined to form seven "component" scores, each with a range of 0-3 points. In all cases, a score of "0" indicates no difficulty and a score of "3" indicates severe difficulty. These seven component scores are then added to yield on "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Held, PhD, Principal Investigator — Queen's University
Locations (1):
- Hydrathletics Inc., Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual IPD among other researchers